CLINICAL TRIAL: NCT04078022
Title: Phase 2b Study of the Safety, Immunogenicity, and Efficacy of a Monovalent Synthetic Carbohydrate-based Conjugate Vaccine (SF2a-TT15) for Protection Against Shigella Flexneri 2a Experimental Infection
Brief Title: Shigella CVD 30000: Study of Responses to Vaccination With Shigella Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Wilbur Chen, MD, MS, Frank M. Calia, MD Endowed Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00086278
Record Dates: First submitted 2019-07-03; First posted 2019-09-04 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Shigella
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Shigella Vaccine or Placebo, Followed by Challenge (Experimental): 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  Interventions: Biological: SF2a-TT15 Shigella Vaccine; Other: Placebo; Biological: S. flexneri 2a strain 2457T Challenge Agent
- Cohort 2: Shigella Vaccine or Placebo, Followed by Challenge (Experimental): 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  Interventions: Biological: SF2a-TT15 Shigella Vaccine; Other: Placebo; Biological: S. flexneri 2a strain 2457T Challenge Agent
- Cohort 3: Shigella Vaccine or Placebo, Followed by Challenge (Experimental): 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  Interventions: Biological: SF2a-TT15 Shigella Vaccine; Other: Placebo; Biological: S. flexneri 2a strain 2457T Challenge Agent
- Cohort 4: Shigella Vaccine Only, No Challenge (Experimental): All volunteers receive the investigational Shigella vaccine (n=12). No Shigella challenge.
  Interventions: Biological: SF2a-TT15 Shigella Vaccine

INTERVENTIONS:
Biological: SF2a-TT15 Shigella Vaccine — 0.5 mL of the vaccine is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
Other: Placebo — 0.5 mL of normal saline is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  Arms: Cohort 1: Shigella Vaccine or Placebo, Followed by Challenge; Cohort 2: Shigella Vaccine or Placebo, Followed by Challenge; Cohort 3: Shigella Vaccine or Placebo, Followed by Challenge
Biological: S. flexneri 2a strain 2457T Challenge Agent — Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
  Arms: Cohort 1: Shigella Vaccine or Placebo, Followed by Challenge; Cohort 2: Shigella Vaccine or Placebo, Followed by Challenge; Cohort 3: Shigella Vaccine or Placebo, Followed by Challenge

SUMMARY:
The purpose of this study is to determine whether SF2a-TT15 (a monovalent synthetic carbohydrate-based conjugate Shigella vaccine) is safe and effective in the prevention of Shigella infection.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether SF2a-TT15 (a monovalent synthetic carbohydrate-based conjugate Shigella vaccine) is safe and effective in the prevention of Shigella infection. This will be a phase 2b, double-blind, placebo-controlled, single-center study, involving a vaccination phase and a challenge phase. The vaccination phase will consist of study participants that will be 1:1 randomized to receive either the vaccine or placebo. Two doses of blinded study product will be given by intramuscular route of administration, separated by approximately 4 weeks. The challenge phase will consist of an inpatient stay of approximately 12 days during which eligible study participants will ingest an oral inoculum of wild-type S flexneri 2a strain 2457T and then be monitored for illness and treated with antibiotics when the primary endpoint is reached or upon 5 days post-challenge, whichever comes first, or when deemed necessary. Upon satisfying discharge criteria, study participants will complete outpatient clinic follow-up visits through ~7 months after last dose of blinded study product (Day 237). The efficacy study will be enrolled through three cohorts of participants, each cohort consisting of approximately 30 subjects that will be involved in the vaccination phase and 22 subjects that will proceed with the challenge phase. There will be a fourth cohort of participants, consisting of 12 subjects, that will receive the vaccine in an open-label design-this cohort will provide serum samples which are intended to be used for generating serum standards for laboratory assays, as a part of ongoing and future clinical development of Shigella vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age 18-45 years
* Provides written informed consent
* Healthy, based on history, exam, and medications
* Documented acceptable screening laboratory work, including:

WBC, ANC, Hg, Platelets Creatinine, ALT, Bili Serum IgA HIV, HBsAg, HCV Negative for HLA-B27 (this criterion does not apply to cohort 4) Stool culture urinalysis

* Passing score on Comprehension Assessment Tool (greater than or equal to 70 percent correct answers)
* Agrees not to participate in another interventional clinical trial during the study period
* For females of child-bearing potential, must agree to acceptable birth control, 4 weeks before enrollment and through 4 weeks after last vaccination or challenge
* Available for a 12-day inpatient stay (this criterion does not apply to cohort 4)

Exclusion Criteria:

* Positive pregnancy test at screening or within 24 hours of study product dosing
* Poor venous access, as defined by inability to obtain venous blood after 3 venipuncture attempts (this criterion does not apply to cohort 4)
* Abnormal vital signs, defined as:

Systolic BP greater than 150 mmHg or Diastolic BP greater than 90 mmHg Resting heart rate greater than 100 Oral temperature greater than or equal to 100.4 degrees F

* Persons with IgA deficiency (serum IgA less than 70 mg per dL
* Serum S. flexneri 2a LPS igG titer greater than or equal to 2500
* Received prior vaccines or had prior infection (natural or challenge) with ETEC or Shigella, within 5 years prior to enrollment
* Symptoms of Traveler's diarrhea associated with travel to countries where Shigella or other enteric infections are endemic (most of the developing world) within 3 years prior to enrollment
* History of chronic gastrointestinal illness, including sever dyspepsia, lactose intolerance, or other significant gastrointestinal tract disease
* Use of antimicrobials within 2 weeks of each dose of vaccine or the challenge
* Regular use (greater than or equal to weekly) of laxatives, anti-diarrheal agents, anti-constipation agents, or antacid therapies
* History of major gastrointestinal surgery (uncomplicated laparoscopic appendectomy or cholecystectomy greater than 1 year prior is permitted)
* Abnormal bowel pattern, defined by less than 3 stools per week or greater than 2 stools per day in the past 6 months
* Use of oral, parenteral or high-dose inhaled steroids within 30 days of each dose of vaccine or the challenge
* Use of any medication which might affect immune function within 30 days of each dose of vaccine or the challenge
* Current medical condition which requires daily or weekly prescribed medications for control (as medication use is limited during the inpatient stay), may be an exclusion criterion if in the judgement of the investigator the potential for missed doses could represent a significant risk to the subject's health
* History of reactive arthritis
* Diagnosis of schizophrenia or other major psychiatric disease
* History of seizure disorder within the last 5 years
* History of alcohol or drug abuse within the last 5 years
* Presence of immunosuppression
* Known significant allergy (i.e., anaphylaxis) to ciprofloxacin, trimethoprim-sulfamethoxazole (Bactrim), or a tetanus-containing vaccine
* 12-lead electrocardiogram with pathologic abnormalities (this criterion does not apply to cohort 4)
* Occupation in food handling industry, living with, or care of very young children (less than 5 years old), elderly (greater than 65 years), or immunocompromised (this criterion does not apply to cohort 4)
* Having any known legal obligations, court appearances, professional meetings, vacations, planned events, or other reasons which might interfere with a person's availability for a 12-day inpatient stay. (this criterion does no apply to cohort 4)
* Any other criteria which, in the investigator's opinion, would compromise the safety of the study, the ability of a subject to participate, or the results of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort 4 was eliminated prior to the start of Cohort 4 enrollment. Cohorts 1-3 are pooled and reported by vaccine vs. placebo recipients.
Groups:
- Shigella Vaccine: 1:1 randomization to investigational Shigella vaccine or placebo (n=29). The majority of participants will then receive the Shigella challenge (n=22).
  SF2a-TT15 Shigella Vaccine: 0.5 mL of the vaccine is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  S. flexneri 2a strain 2457T Challenge Agent: Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
- Placebo: 1:1 randomization to investigational Shigella vaccine or placebo (n=29). The majority of participants will then receive the Shigella challenge (n=22).
  Placebo: 0.5 mL of normal saline is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  S. flexneri 2a strain 2457T Challenge Agent: Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
Period: Vaccination Phase
Arm/Group | Shigella Vaccine | Placebo
Started | 29 | 29
Completed | 27 | 26
Not Completed | 2 | 3
Not completed — Withdrawal prior to challenge | 2 | 3
Period: Challenge Phase
Arm/Group | Shigella Vaccine | Placebo
Started | 22 | 22
Completed | 21 | 22
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vaccine: 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  SF2a-TT15 Shigella Vaccine: 0.5 mL of the vaccine is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
- Placebo: 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  Placebo: 0.5 mL of normal saline is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 32 [20 to 44] | 32 [20 to 45] | 32 [20 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 14 | 19 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 20 | 20 | 40
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate-Severe Shigellosis Illness, With Challenge
Description: Count of participants with primary endpoint (Moderate-Severe Shigellosis)
Time Frame: 10 days after challenge
Population: All participants that were randomized to vaccine or placebo and were challenged
Measure: Count of Participants; unit: Participants
Groups:
- Shigella Vaccine: 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  SF2a-TT15 Shigella Vaccine: 0.5 mL of the vaccine is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  S. flexneri 2a strain 2457T Challenge Agent: Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
- Placebo: 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  Placebo: 0.5 mL of normal saline is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  S. flexneri 2a strain 2457T Challenge Agent: Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
Arm/Group | Shigella Vaccine | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 14 | 17

2. Secondary Outcome: Number of Participants Meeting Other Case Definitions and Endpoint Definitions
Time Frame: 10 days after challenge
Population: Participants randomized to vaccine or placebo and were challenged
Measure: Count of Participants; unit: Participants
Arm/Group | Shigella Vaccine | Placebo
Number analyzed (Participants) | 22 | 22
Participants
  Count of participants with any diarrhea endpoint | 15 | 18
  Count of participants with any dysentery endpoint | 4 | 12
  Count of participants with any fever endpoint | 12 | 15
  Count of participants with any combination of diarrhea, dysentery, and/or fever | 16 | 19

3. Secondary Outcome: Number of Participants With Anti-LPS Serum IgG ELISA Response
Description: Anti-LPS serum IgG ELISA response, by response rates (proportion of 4-fold increases from baseline, Day 1)
Time Frame: Days 29, 57 and 85
Population: Enrolled participants
Measure: Count of Participants; unit: Participants
Groups:
- Vaccine Enrolled; Vaccine Challenged: 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  SF2a-TT15 Shigella Vaccine: 0.5 mL of the vaccine is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  S. flexneri 2a strain 2457T Challenge Agent: Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
- Placebo Enrolled; Placebo Challenged: 1:1 randomization to investigational Shigella vaccine or placebo (n=30). The majority of participants will then receive the Shigella challenge (n=22).
  Placebo: 0.5 mL of normal saline is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  S. flexneri 2a strain 2457T Challenge Agent: Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
Arm/Group | Vaccine Enrolled | Placebo Enrolled | Vaccine Challenged | Placebo Challenged
Number analyzed (Participants) | 29 | 29 | 22 | 22
Participants
  Count of participants with serum IgG ELISA response rates, post-dose 1 (Day 29) | 27 | 1 | 20 | 1
  Count of participants with serum IgG ELISA response rates, post-dose 2 (Day 57) | 26 | 1 | 21 | 1
  Count of participants with serum IgG ELISA response rates, post-challenge (Day 85) | 26 | 17 | 22 | 17

4. Secondary Outcome: Anti-LPS Serum IgG ELISA Response, by Titer
Time Frame: Days 1, 29, 57 and 85
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Vaccine Enrolled | Placebo Enrolled | Vaccine Challenged | Placebo Challenged
Number analyzed (Participants) | 29 | 29 | 22 | 22
titer
  Mean ±SD pre-vaccination (Day 1) | 1020.69 (1143.11) | 662.07 (638.87) | 800 (489.9) | 772.73 (696.37)
  Mean ±SD post-dose 1 (Day 29) | 17441.38 (21018.59) | 965.52 (1549.03) | 18190.91 (22253.3) | 1172.73 (1734.02)
  Mean ±SD post-dose 2 (Day 57) | 15318.52 (13574.1) | 965.38 (1285.91) | 16327.27 (14392.93) | 1081.82 (1368.57)
  Mean ±SD post-challenge (Day 85) | 18755.56 (14338.9) | 5850 (6204.14) | 21345.45 (14537.76) | 6940 (6251.27)

5. Secondary Outcome: Serum Bactericidal Activity Response, by Response Rates (Proportion of 4-fold Increases From Baseline, Day 1)
Time Frame: Days 29, 57 and 85
Population: Enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Enrolled | Placebo Enrolled | Vaccine Challenged | Placebo Challenged
Number analyzed (Participants) | 29 | 29 | 22 | 22
Participants
  Count post-dose 1 (Day 29) | 21 | 2 | 17 | 2
  Count post-dose 2 (Day 57) | 22 | 1 | 17 | 1
  Count post-challenge (Day 85) | 23 | 12 | 19 | 12

6. Secondary Outcome: Serum Bactericidal Activity Response, by Titer
Time Frame: Days 1, 29, 57 and 85
Population: Enrolled participants
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Vaccine Enrolled | Placebo Enrolled | Vaccine Challenged | Placebo Challenged
Number analyzed (Participants) | 29 | 29 | 22 | 22
titer
  Mean ±SD pre-vaccination (Day 1) | 1131.48 (2542.76) | 399.04 (723.1) | 1229.55 (2752.74) | 279.55 (466.6)
  Mean ±SD post-dose 1 (Day 29) | 11973.15 (38813.69) | 1856.73 (5465.05) | 13729.55 (42920.28) | 2006.82 (5923.36)
  Mean ±SD post-dose 2 (Day 57) | 8553.7 (19417.73) | 745.19 (1723.18) | 9147.73 (21379.99) | 547.73 (1388.06)
  Mean ±SD post-challenge (Day 85) | 8479.63 (19301.06) | 2345.83 (3228.33) | 9420.45 (21232.07) | 2448.75 (3326.45)

ADVERSE EVENTS:
Time Frame: The assessment of the safety of the vaccine was through the detection and documentation of adverse effects, both solicited AEs and unsolicited AEs, and/or clinically significant laboratory abnormalities, from enrollment through 28 days post-vaccination. Only the occurrence of SAEs were reported between Day 57 (or 28 days post-last dose of vaccine) through the end of the study (Day 237).
Groups:
- Vaccine Enrolled: 1:1 randomization to investigational Shigella vaccine or placebo (n=29). The majority of participants will then receive the Shigella challenge (n=22).
  SF2a-TT15 Shigella Vaccine: 0.5 mL of the vaccine is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  S. flexneri 2a strain 2457T Challenge Agent: Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
- Placebo Enrolled; Vaccine Challenged; Placebo Challenged: 1:1 randomization to investigational Shigella vaccine or placebo (n=29). The majority of participants will then receive the Shigella challenge (n=22).
  Placebo: 0.5 mL of normal saline is administered via an intramuscular injection into the deltoid muscle on Study Day 1 and Study Day 29.
  S. flexneri 2a strain 2457T Challenge Agent: Each participant will drink 120 mL of sodium bicarbonate buffer solution. Approximately 1 to 2 minutes later, the participant will ingest approximately 1500 cfu of S. flexneri 2a strain 2457T suspended in 30 mL of the bicarbonate buffer solution.
Arm/Group | Vaccine Enrolled | Placebo Enrolled | Vaccine Challenged | Placebo Challenged
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 18/29 | 21/29 | 0/22 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine Enrolled (N=29) | Placebo Enrolled (N=29) | Vaccine Challenged (N=22) | Placebo Challenged (N=22)
Syncope (Cardiac disorders) | 1 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 0
Injection Site Pain (General disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Facial Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0
Bilirubin Increased (Investigations) | 0 | 3 | 0 | 0
Blood Pressure Decreased (Investigations) | 0 | 1 | 0 | 0
Blood Pressure Diastolic Increased (Investigations) | 1 | 0 | 0 | 0
Blood Pressure Systolic Increased (Investigations) | 1 | 0 | 0 | 0
Heart Rate Increased (Investigations) | 1 | 3 | 0 | 0
Hemoglobin Decreased (Investigations) | 1 | 0 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0
White Blood Cell Count Increaed (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Foot Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Wrist Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Burn (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT04078022/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT04078022/SAP_001.pdf